CLINICAL TRIAL: NCT06884891
Title: A Multicenter Randomized, Double-blinded, Parallel, Positive-controlled, Phase Ⅲ Comparative Study to Evaluate the Efficacy and Safety of QL2108 to Dupixent® in Adult Subjects With Moderate-to-Severe Atopic Dermatitis.
Brief Title: A Phase Ⅲ Comparative Study of QL2108 to Dupixent®
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL2108-301
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2108 injection (Experimental): QL2108 injection; 300mg/2.0mL; subcutaneous injection
  Interventions: Drug: QL2108 injection
- Dupixent® (Active Comparator): Dupixent®; 300mg/2.0mL; subcutaneous injection
  Interventions: Drug: Dupixent®

INTERVENTIONS:
Drug: QL2108 injection — 300mg/2.0mL; an initial dose of 600 mg (two 300 mg injections), followed by 300 mg given every other week (Q2W);subcutaneous injection
  Arms: QL2108 injection
Drug: Dupixent® — 300mg/2.0mL; an initial dose of 600 mg (two 300 mg injections), followed by 300 mg given every other week (Q2W); subcutaneous injection
  Arms: Dupixent®

SUMMARY:
It is a multicenter randomized, double-blinded, parallel, positive-controlled, Phase Ⅲ comparative study to evaluate the efficacy and safety of QL2108 to Dupixent® in adult subjects with moderate-to-severe atopic dermatitis. A total of 520 subjects are planned to be included and randomized at a ratio of 1:1 to receive QL2108 injection or Dupixent®

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged from 18 to 75 years (including the boundary value)
* At the time of screening, the diagnosis of atopic dermatitis (AD) meets the Hanifin-Rajka criteria, with a disease history of ≥1 year prior to screening.
* During the screening period and prior to randomization: EASI score ≥16, IGA score ≥3, BSA ≥10%.

Exclusion Criteria:

* People who have previously used or participated in clinical trials of monoclonal antibody with the same target or dupilumab
* Having participated in drug or device clinical trials within 12 weeks or 5 half-lives of other investigational drugs before the study administration.
* Subjects who have received live vaccines or live-attenuated vaccines within 12 weeks prior to randomization or plan to receive such vaccines during the trial period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving EASI-75 at week 16. | 16 weeks
  EASI-75

SECONDARY OUTCOMES:
Proportion of patients achieving EASI-75 at week 52 | 52 weeks
  EASI-75
Proportion of patients achieving IGA-TS (IGA score was 0 or 1 and decreased by ≥2 points from baseline) at week 16 and week 52 | 16 weeks and 52 weeks
  IGA-TS